CLINICAL TRIAL: NCT04623827
Title: A Retrospective Study Concerning the Psycho-attitudinal Classification of Patients Suffering From Fibromyalgia Undergoing a Specialized Analgesic Treatment
Brief Title: Retrospective Study of Psychoattitudinal Patterns in Patients With Fibromyalgia Receiving Antalgic Therapy
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Andrea Fanelli, Principal Investigator, University of Bologna
Other Study IDs: FIBRO_PATTERN
Record Dates: First submitted 2020-09-19; First posted 2020-11-10 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Analgesia; Fibromyalgia; Pain, Chronic; Pain Syndrome
Keywords: Fibromyalgia; Pain, Chronic; Analgesia
MeSH Terms: conditions — Agnosia; Fibromyalgia; Chronic Pain; Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fibromyalgia (FM) is a widespread and invalidating disease that requires a multidisciplinary approach. Particularly, the psychiatric component seems to influence the algological management of these patients. Since January 2018, the HADS, SF-36, IMSA, TCI psycho-attitudinal questionnaires have been introduced in the Pain Therapy unit of Policlinico Sant'Orsola-Malpighi in an attempt to improve the care of patients diagnosed with FM.

The aim of the study is to identify, through retrospective evaluation of TCI tests and its subdomains, compiled by patients with FM diagnosis, Pain Avoidance and Pain Persistance personality patterns, indicated in the literature. Anxiety and Depression incidence is also observed through retrospective evaluation of HADS tests.

Patients in the Antalgic Therapy Outpatient Clinic diagnosed with FM, aged ≥18 years, who have completed selfadministered psychoattitudinal tests from January 2018 to January 2019 were considered. The data were collected in aggregate and extrapolated anonymously.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia
* years ≥ 18

Exclusion Criteria:

* not present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of fibromyalgia who come to the pain therapy service over the age of 18 between January 2018 and January 2019..
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Psycho-attitudinal Pattern | 1 year
  A retrospective evaluation of the Temperament and Character Inventory test scores in the period from January 2018 to January 2019 by patients diagnosed with Fibromyalgia related to the antalgic therapy clinic.

SECONDARY OUTCOMES:
Anxiety and depression | 1 year
  To investigate the presence of moderate to severe anxiety-depressive disorders among patients with anxiety and depression at the antalgic therapy clinic using the HADS tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Fanelli, Bologna, Italy